CLINICAL TRIAL: NCT04728750
Title: Laparoscopic Enucleation of Frantz's Tumor of the Pancreas: Case Report and Literature Review
Brief Title: Laparoscopic Enucleation of Frantz's Tumor of the Pancreas
Status: Completed | Type: Observational
Sponsor: Tecnologico de Monterrey (Other)
Responsible Party: Principal Investigator, Alejandro Ruiz Velasco Santacruz, Clinical Professor, Tecnologico de Monterrey
Other Study IDs: FT7831
Record Dates: First submitted 2021-01-21; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Solid Pseudopapillary Neoplasm of the Pancreas

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Enucleation of a tumor of the pancreas — Enucleation of a tumor in the pancreas is feasible and safe, as it offers a minimally invasive approach, and morbidities are fewer than open or conventional approach

SUMMARY:
The present study describes a 32-year-old female patient, in whom a preoperative imaging diagnosis confirmed a mass in the junction of the body and tail of the pancreas. Based on the anamnesis, on the preoperative diagnosis, and on the general status of the patient, the decision was made to performed laparoscopic enucleation of the pancreatic tumor. The operation and postoperative recovery passed without complications. A minimally invasive surgical approach should be applied whenever the dimensions and the localization of the tumor permits it, bearing in mind all the benefits and advantages that this surgical technique has to offer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with benign tumor of the pancreas
* Patients with a size tumor of less than 3 cm on the pancreas

Exclusion Criteria:

* Patients with a size tumor greater than 3 cm on the pancreas
* Malignant tumors of the pancreas

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosed pancreatic tumor by image study.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-02 (Actual)

PRIMARY OUTCOMES:
Complete enucleation of a tumor in the pancreas | December 2020
  Performance of a laparoscopic enucleation of a tumor in the pancreas, and compared it with a conventional approach

CONTACTS AND LOCATIONS:
Locations (1):
- Escuela Nacional de Medicina, Tecnologico de Monterrey, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No